CLINICAL TRIAL: NCT04853329
Title: Phase 1/2, Multicenter, First-In-Human, Dose Escalation and Dose Expansion Study of CPO107 Administered Intravenously to Patients with Advanced CD20-positive Non-Hodgkins Lymphoma
Brief Title: Dose Escalation and Expansion Study of CPO107 for Patients with Advanced CD20-positive Non-Hodgkins Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Conjupro Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPO107-US-1001
Record Dates: First submitted 2021-03-02; First posted 2021-04-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: CD20 Positive Non Hodgkin Lymphoma
Keywords: CD20 positive; Non Hodgkin Lymphoma; CD20 CD47; CPO107; Phase 1/2
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- PartA- Arm A (Experimental): Arm A 1-6 subjects will be enrolled at dose levels of CPO107 at (1, 3, 6, 12, 20 mg/kg).
  Each subject group will receive multiple cycles of a weekly dose of CPO-107 (1 cycle=21 days=3 treatments).
  Interventions: Drug: CPO107
- PartA- Arm B (Experimental): Arm B will explore a 3 weekly schedule in which a single dose is administered every 3 weeks (1 cycle=21 days=1 treatment). The starting dose for Arm B will be the dose level below the Arm A level that provides an equivalent dose over a 3-week period.
  Interventions: Drug: CPO107
- Part B (Experimental): Part B with either: second or greater relapse OR refractory patients, as defined by not achieving a CR after 2 cycles of a standard first line chemoimmunotherapy regimen or not achieving a CR following 1 cycle of a second line chemotherapy regimen.
  Interventions: Drug: CPO107

INTERVENTIONS:
Drug: CPO107 — CD20-CD47 Bispecific Fusion Protein
  Other Names: JMT601

SUMMARY:
This first-in-human Phase 1 study will be a multicenter, dose-escalating, single-agent study conducted in patients with advanced CD20-associated hematological cancers for which the investigator determines there to be no other higher priority therapies available.

DETAILED DESCRIPTION:
This first-in-human Phase 1 study will be a multicenter, dose-escalating, single-agent study conducted in patients with advanced CD20-associated hematological cancers for which the investigator determines there to be no other higher priority therapies available. All patients must have failed at least two prior lines of conventional systemic therapy that must also include an approved CD20 based treatment. All patients will need to have CD20-positive disease, as determined by the expression of CD20 on tumor cells assayed within 6 months prior to study entry.

The study will consist of 2 parts, Part A and Part B. In Part A of the study, dose escalation will proceed according to the guidelines in the Treatment and Dosing section below, following a rule-based design methodology. Two different schedules will be explored to establish the PK profile and thus better inform the selection of the final dosing schedule to be developed. Arm A will explore a continuous weekly dosing schedule and will commence first. Arm B will explore a 3 weekly schedule in which a single dose is administered every 3 weeks. Part B dose expansion of the study will commence, in which a single dosing schedule will be explored in CD20-positive patients. The schedule will be selected based on PK and safety determinants from Study Part A.

ELIGIBILITY:
Inclusion Criteria:

The following key inclusion criteria apply to both Part A and Part B:

* Diagnosis of CD20 positive NHL. CD20 assay to have been performed within 6 months prior to protocol entry. Eligible NHL subtypes include Diffuse Large B-Cell Lymphoma (DLBCL, not otherwise specified, NOS), Follicular Lymphoma, Chronic lymphocytic leukemia/small lymphocytic lymphoma, B cell prolymphocytic leukemia and Mantle cell lymphoma.
* Patients with SLL must have received, or not be eligible for, BTK and BCL-2 inhibitor therapy.
* Disease progression or relapse following at least two prior lines of conventional systemic therapy for advanced disease. Dosing regimen must have included a CD20 targeted therapy (for example, RCHOP).
* A clinical indication for treatment must be present for patients with Follicular Lymphoma and Chronic/Small/Prolymphocytic/Mantle B-cell non-Hodgkin lymphoma.
* Having at least one measurable target lesion present and documented by RECIST 1.1.
* Adequate organ function, such as Renal function, Hepatic Function, Cardiovascular, Adequate hematological reserve.
* Complete resolution of all prior toxicities from prior anticancer therapy, defined as having resolved to baseline or to common terminology criteria for adverse events (CTCAE) grade≤1, with the exception of alopecia, or to the levels dictated in the inclusion/exclusion criteria, and a washout period of 5 half-lives of prior small molecule systemic therapy.
* Life expectancy >12 weeks.
* Age: Lower age limit of 18 years.
* ECOG performance status 0 or 1 at screening.
* Ability to understand the nature of this study, comply with protocol requirements, and give written informed consent. For minors, legal guardian willingness to give written informed consent with patient assent, where appropriate.
* Patients of reproductive potential: All female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before study entry.

Exclusion Criteria:

The following key exclusion criteria apply:

* Patients with indolent Follicular Lymphoma or Chronic/Small/Prolymphocytic/Mantle B-cell non-Hodgkin lymphoma in need of immediate cytoreductive therapy are excluded, unless the patient has no remaining treatment choice with potential benefit.
* Patient has participated in any investigational research study and is being screened for participation within a period of 5 half-lives, or 4 weeks of the last dose of the investigational therapy, whichever is longer.
* Patients with history of severe hypersensitivity reactions to anti-CD20 treatment or any components of study drug formulation.
* Presence or recent history within 6 months of arteritis or any systemic clotting disorder, thrombotic or thromboembolic events.
* History or presence of autoimmune conditions; patients who have a medical condition that requires chronic systemic steroid therapy or requires any other form of immunosuppressive medication.
* Patients with a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >480 milliseconds (ms) (CTCAE grade 1) using Fredericia's QT correction formula.
* Active or latent hepatitis B or active hepatitis C or any uncontrolled infection at screening; HIV positive test within 8 weeks of screening.
* Serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
* Presence of other active cancers, or history of treatment for invasive cancer ≤3 years.
* Patients who started erythropoietin or granulocyte colony-stimulating factor (G-CSF), pegfilgrastim, or filgrastim ≤4 weeks prior to the first dose of the study drug.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Active CNS disease involvement; CNS directed radiation must be completed >8 weeks prior to CPO107 infusion.
* Non-CNS site of radiation must be completed >2 weeks prior to CPO107 infusion.
* Pregnant or nursing (lactating) women
* And others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
To determine the recommended single-agent CPO107 RP2D | through study completion, an average of 1 year
  To determine the recommended single-agent CPO107 RP2D and schedule for further exploration in CD20 positive Non-Hodgkins Lymphoma.

SECONDARY OUTCOMES:
Safety assessment-Incidence of treatment-emergent AEs (TEAEs) | through study completion, an average of 1 year
  Safety will be assessed through the analysis of the reported incidence of treatment-emergent AEs (TEAEs) by evaluating adverse events based on laboratory results, vital signs and ECG findings.
Pharmacokinetic (PK) | through study completion, an average of 1 year
  The pharmacokinetic of CPO-107 will be assessed by measuring the blood concentration of the drug in the plasma at various timepoints and calculation of parameters, such as Peak Plasma Concentration (Cmax).
Expression of anti-drug antibody (ADA) | through study completion, an average of 1 year
  The expression of anti-drug antibodies (ADAs) following administration will be assessed by analysis of serum samples.
Efficacy assessment | through study completion, an average of 1 year
  To document any early indication of clinical efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Novick, MD PhD, Study Director — Conjupro Biotherapeutics, Inc.
Locations (1):
- Novant Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Undecided